CLINICAL TRIAL: NCT04922749
Title: Evaluation of the Implementation and Effectiveness of a Multidisciplinary Lifestyle Treatment for Inpatients With Mental Illness (MULTI+)
Brief Title: Evaluation of a Multidisciplinary Lifestyle Treatment for Inpatients With Mental Illness
Acronym: MULTI+
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: GGZ Centraal (Other)
Collaborators: Stichting tot steun VCVGZ (Other); UMC Utrecht (Other); Maastricht University (Other); The Healthcare Innovation Centre (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 200333; 277 (Other Grant/Funding Number: Stichting tot steun VCVGZ)
Record Dates: First submitted 2021-06-03; First posted 2021-06-11 (Actual); Last update posted 2021-11-16 (Actual); Status verified 2021-06

CONDITIONS: Mental Illness; Lifestyle
Keywords: Inpatients; Implementation
MeSH Terms: conditions — Mental Disorders

STUDY DESIGN:
Intervention Model Description: Prospective open cohort stepped wedge cluster randomized trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TAU (No Intervention): Treatment as usual (TAU); consist mainly of pharmacological treatment and psychotherapy.
- MULTI+ (Experimental): Lifestyle treatment
  Interventions: Behavioral: MULTI+

INTERVENTIONS:
Behavioral: MULTI+ — MULTI+ is a multidisciplinary, multicomponent treatment which aims to improve lifestyle factors through a holistic lifestyle approach, by focusing on 10 core components. The MULTI+ will be integrated into daily treatment to promote uptake and sustainability.
  Arms: MULTI+

SUMMARY:
People with mental illness (MI) have a reduced life expectancy compared to the general population, mostly attributable to somatic diseases caused by poor physical health. Modifiable "lifestyle factors" have been increasingly associated with the onset of somatic diseases in people with MI and refer to health behaviours such as physical activity (PA), diet, sleep and smoking behaviour. Despite the evidence demonstrating the efficacy of interventions aimed at improving lifestyle factors, there have not been many structural changes in routine clinical care for people with MI. Using a multidisciplinary, multicomponent approach, Deenik and colleagues (2019) were the first to find long-term positive effects in both mental and somatic health in a real-world inpatient setting for people with severe mental illness (SMI). They found improvements in metabolic health, psychosocial functioning and quality of life, and a reduction in the use of psychotropic medication. The authors urged to confirm and complement findings in scaled-up studies, and made several suggestions for improvement of the treatment and pragmatic research of implementation. In line with these previous recommendations the MULTI is being scaled-up into the MULTI+. This study investigates the implementation and effectiveness of a multidisciplinary lifestyle treatment for inpatients with mental illness (MULTI+).

DETAILED DESCRIPTION:
Study design and setting

This study is a prospective open cohort stepped wedge cluster randomized trial with continuous recruitment. This study is being conducted at the inpatient psychiatric wards, covering approximately 750 places of residency in which approximately 2000 patients are treated annually, from the specialist mental healthcare organisation GGz Centraal (the Netherlands). The study uses a stepped-wedge clustered design. The psychiatric wards are divided into three clusters, based on their geographical locations. These clusters gradually implement MULTI+ in semi-annual steps, such that all clusters are exposed to the MULTI+ at the end of the study. The repeated measurements are conducted on ward-level, rather than individual patient level.

Intervention

MULTI+ is a multidisciplinary, multicomponent treatment which aims to improve lifestyle factors through a holistic lifestyle approach, by focusing on 10 core components. Core components refer to essential elements and activities that are necessary to achieve desired outcomes. The core components of MULTI+ are based on previous recommendations and existing literature. The core components of MULTI+ are routine daily structure and sleep, physical activity, attention to nutrition and eating habits, smoking cessation, multidisciplinary treatment, skills training, psychoeducation, critical review of obesogenic environment and existing policies, active participation of health care professionals (HCPs), and training of HCPs. The core components are co-designed and tailored to the ward and patient population, because of the large heterogeneity in patient characteristics and varying access to facilities and staffing.

Analyses

To measure the intervention effect, linear mixed models will be used for continuous outcome measures and logistic mixed models for dichotomous outcome measures. In each model, the intervention effect will be estimated as the difference between the postintervention and preintervention levels of the outcome after adjusting for time as a categorical variable. All models will be corrected for group differences at baseline and the baseline differences of the outcome measures concerned (to account for regression to the mean).

ELIGIBILITY:
Inclusion Criteria:

* 16 years or older
* Mentally ill inpatients
* Receive care at the inpatient psychiatric wards of GGz Centraal where the MULTI+ will be implemented

Exclusion Criteria:

* Limited knowledge or understanding of Dutch
* If their psychiatric or physical condition hinders informed consent at the discretion of the relevant physician, nurses, or researcher

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 846 (Estimated)
Dates: Start 2020-07-01 (Actual); Primary Completion 2022-09-01 (Estimated); Study Completion 2022-09-01 (Estimated)

PRIMARY OUTCOMES:
QRISK3 score | 4 measurements semi-annually over a period of 24 months
  Algorithm that estimates the probability of developing cardiovascular disease over the next 10 years by taking multiple risk factors into account.

SECONDARY OUTCOMES:
Change in metabolic health: Waist circumference | 4 measurements semi-annually over a period of 24 months
  waist circumference measured halfway between the iliac crest and lowest rib in standing position
Change in metabolic health: Systolic and diastolic blood pressure | 4 measurements semi-annually over a period of 24 months
  Measured systolic and diastolic blood pressure (mmHg)
Change in metabolic Health:Lipids | 4 measurements semi-annually over a period of 24 months
  Values in blood sample
Change in metabolic Health: HDL Cholesterol | 4 measurements semi-annually over a period of 24 months
  Values in blood sample
Change in metabolic Health: triglycerides | 4 measurements semi-annually over a period of 24 months
  Values in blood sample
Change in metabolic Health: Fasting glucose | 4 measurements semi-annually over a period of 24 months
  Values in blood sample
Weight Change | 4 measurements semi-annually over a period of 24 months
  Weight is measured to the nearest 0.1 kg.
Change in BMI | 4 measurements semi-annually over a period of 24 months
  weight divided by height in meters squared
Change in medication use through daily defined doses (DDD) | 4 measurements semi-annually over a period of 24 months
  Medication prescribed for cardiovascular health and diabetes, and psychotropic medication will be converted into daily defined doses (DDD) according the Anatomical Therapeutic Chemical Classification System from the World Health Organization (WHO). Medication data is obtained from patient files.
Change in psychosocial functioning: Adults | 4 measurements semi-annually over a period of 24 months
  Measured by the Health of the Nations Outcomes Scale (HoNOS-12). All items are scored on a 5-point Likert scale, ranging from 0 (no problem) to 4 (severe problem).
Change in psychosocial functioning: Elderly | 4 measurements semi-annually over a period of 24 months
  Measured by the Health of the Nations Outcomes Scale (HoNOS-65+). All items are scored on a 5-point Likert scale, ranging from 0 (no problem) to 4 (severe problem).
Change in psychosocial functioning: Adolescents | 4 measurements semi-annually over a period of 24 months
  Measured by the Health of the Nations Outcomes Scale (HoNOSCA). All items are scored on a 5-point Likert scale, ranging from 0 (no problem) to 4 (severe problem).
Change in substance use | 4 measurements semi-annually over a period of 24 months
  Measured by routine questions about smoking, alcohol use and soft drugs
Change in diet | 4 measurements semi-annually over a period of 24 months
  Measured by a 24-hour dietary recall (24HR)
Change in dietary habits | 4 measurements semi-annually over a period of 24 months
  Measured by the Three Factor Eating Questionnaire Revised 18-items (TFEQ-R18), which consists of 18 items on a 4 point measuring scale, measuring cognitive restraint, uncontrolled eating and emotional eating. Raw scale scores are transformed on a scale from 0-100 (raw score- lowest possible score/possible raw score range)*100).
Change in physical activity (PA): PaVs | 4 measurements semi-annually over a period of 24 months
  Measured by the physical activity vital sign (PaVs). The PaVs is a two-item questionnaire, recommended as a brief way to routinely gain insight in physical activity levels. The PaVs can be used to assess whether the national activity guideline for aerobic activity are met in the context of health considerations (yes = 1, no = 0). Higher score means that the national activity guidelines are met.
Change in physical activity (PA): SIMPAQ | 4 measurements semi-annually over a period of 24 months
  Measure by the Simple Physical activity Questionnaire (SIMPAQ). The SIMPAQ consists of five items (boxes), and participants are asked about time spent in bed (box 1), time sedentary, including naps (box 2), time spent walking (box 3), time spent exercising (box 4) and time spent in incidental activity, such as housekeeping (box 5). The total self-reported time spent on moderate-vigorous physical activity (MVPA) can be calculated by adding box 4 and 5.
Change in sleep (SCOPA-sleep) | 4 measurements semi-annually over a period of 24 months
  Measured by the Scales for Outcomes in Parkinson's Disease - Sleep (SCOPA-Sleep). The SCOPA-Sleep is developed to evaluate night-time sleep and daytime sleepiness in a short and practical manner. The questionnaire enquires about the use of sleep medication and if so, which medication. It then uses 5 items to evaluate night-time sleep, 1 question inquiring overall quality of sleep followed by 6 items to evaluate daytime sleepiness on a 4 point Likert scale ranging from 0 (not at all) to 4 (a lot).
Change in psychopathology (BSI) | 4 measurements semi-annually over a period of 24 months
  Measured by the Brief Symptom Inventory (BSI). The BSI comprises 53 items that reflect 9 symptom domains of psychopathology (somatization, obsessive compulsive, interpersonal sensitivity, depression, anxiety, hostility, phobic anxiety, paranoid ideation and psychoticism). Each item is rated on a 5-point scale of distress from 0 (not at all) to 4 (extremely).
Change in Quality of life (WHOQoL-Bref) | 4 measurements semi-annually over a period of 24 months
  Measured by the World Health Organisation Quality of Life-BREF (WHOQoL-BREF). The four WHOQoL-BREF domains are measured through 24 domain-specific items: Physical health (7 items), Psychological (6 items), Social relations (3 items) and Environment (8 items) and two general health items. Item scores have various options but always range from 1 to 5, such as very poor to very good or not at all to extremely, and will be converted to domain scores (range from 4 to 20) based on the WHO guidelines. Higher score reflect a better quality of life.
Change in Quality of life (EQ-5D) | 4 measurements semi-annually over a period of 24 months
  Measured by the EuroQol 5D (EQ-5D).The EQ-5D is a generic instrument that consists of 5 dimensions of health, with one item per dimension; mobility, selfcare, usual activities, pain/discomfort, and anxiety/depression. There are three levels of severity ranging from no issues to many issues. The index score are calculated ranging from 0 (worst quality of life) to 1 (perfect quality of life).
Change in meaning in life (MHC-SF) | 4 measurements semi-annually over a period of 24 months
  Measured by the Mental Health Continuum - Short Form (MHC-SF). The MHC-SF measures positive mental health and consists of 14 items, representing feelings of well-being: Emotional well-being (three items), Psychological well-being (six items), and Social well-being (five items). Participants rate the frequency of these feelings in the past month on a 6-point Likert scale (never, once or twice a month, about once a week, two or three times a week, almost every day, every day).
Barriers and facilitators of the implementation of the MULTI+ (MIDI) | 4 measurements semi-annually over a period of 24 months
  Measured by the Measurement Instrument for Determinants of the Innovation (MIDI). The MIDI is comprised of 28 items, divided into 4 scales measuring determinants associated with innovations (7 items), the user (11 items) and the organization (10 items). All items are scored on a 5-point Likert scale ranging from 1 (totally disagree) to 5 (totally agree). Items which ≥20% responds negatively (disagree/totally disagree) are considered barriers. Items which ≥80% respond positively (agree/totally agree) are considered facilitators.
Change in amount of adverse events | 24 months
  Institutional software in which employees register and categorize adverse events (e.g. aggression).
Change in motivation for behavioural regulation for physical activity | 4 measurements semi-annually over a period of 24 months
  Measured by the Behavioural Regulation in Exercise Questionnaire (BREQ-2). The BREQ-2 is comprised of 19 items, divided into 5 scales measuring; Amotivation (item 5, 9 12, 19), External (item 1, 6, 11, 16), Identified (item 2, 7, 13), Introjected (item 3, 8, 14, 17), and Intrinsic (item 4, 10, 15, 18 ) regulations. The mean scores for each scale can be used as a multidimensional instrument, giving separate scores for each subscale.
Change in motivation for behavioural regulation for healthy diet | 4 measurements semi-annually over a period of 24 months
  Based on the BREQ-2 as used in this study, the researchers devised a behavioural regulation diet questionnaire. All mentioning of "exercise" in the BREQ-2 has been replaced by referring to "(eat a) healthy diet". This questionnaire comprised of 19 items, divided into 5 scales measuring; Amotivation (item 5, 9 12, 19), External (item 1, 6, 11, 16), Identified (item 2, 7, 13), Introjected (item 3, 8, 14, 17), and Intrinsic (item 4, 10, 15, 18 ) regulations. The mean scores for each scale can be used as a multidimensional instrument, giving separate scores for each subscale.
Health Technology Assessment (HTA) | 24 months
  Cost-effectiveness will be investigated through calculation of the costs of treatment as usual as compared to costs of MULTI+

OTHER OUTCOMES:
Process evaluation - Change in RE-AIM domains | 24 months
  The process evaluation is conducted using the RE-AIM framework (RE-AIM). Reach, Efficacy, Adoption, Implementation and Maintenance will be assessed continuously throughout the study. There are no scores attached to the domains, rather, change is evaluated.

CONTACTS AND LOCATIONS:
Locations (1):
- GGz Centraal, Amersfoort, Utrecht, Netherlands

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hjorthoj C, Sturup AE, McGrath JJ, Nordentoft M. Years of potential life lost and life expectancy in schizophrenia: a systematic review and meta-analysis. Lancet Psychiatry. 2017 Apr;4(4):295-301. doi: 10.1016/S2215-0366(17)30078-0. Epub 2017 Feb 22. PMID 28237639
- [Background] Correll CU, Solmi M, Veronese N, Bortolato B, Rosson S, Santonastaso P, Thapa-Chhetri N, Fornaro M, Gallicchio D, Collantoni E, Pigato G, Favaro A, Monaco F, Kohler C, Vancampfort D, Ward PB, Gaughran F, Carvalho AF, Stubbs B. Prevalence, incidence and mortality from cardiovascular disease in patients with pooled and specific severe mental illness: a large-scale meta-analysis of 3,211,768 patients and 113,383,368 controls. World Psychiatry. 2017 Jun;16(2):163-180. doi: 10.1002/wps.20420. PMID 28498599
- [Background] Deenik J, Czosnek L, Teasdale SB, Stubbs B, Firth J, Schuch FB, Tenback DE, van Harten PN, Tak ECPM, Lederman O, Ward PB, Hendriksen IJM, Vancampfort D, Rosenbaum S. From impact factors to real impact: translating evidence on lifestyle interventions into routine mental health care. Transl Behav Med. 2020 Oct 8;10(4):1070-1073. doi: 10.1093/tbm/ibz067. PMID 31169897
- [Background] Deenik J, Tenback DE, Tak ECPM, Hendriksen IJM, van Harten PN. [Thinking inside the box: improving the lifestyle of inpatients with severe mental illness]. Tijdschr Psychiatr. 2020;62(7):564-574. Dutch. PMID 32700302
- [Background] Firth J, Siddiqi N, Koyanagi A, Siskind D, Rosenbaum S, Galletly C, Allan S, Caneo C, Carney R, Carvalho AF, Chatterton ML, Correll CU, Curtis J, Gaughran F, Heald A, Hoare E, Jackson SE, Kisely S, Lovell K, Maj M, McGorry PD, Mihalopoulos C, Myles H, O'Donoghue B, Pillinger T, Sarris J, Schuch FB, Shiers D, Smith L, Solmi M, Suetani S, Taylor J, Teasdale SB, Thornicroft G, Torous J, Usherwood T, Vancampfort D, Veronese N, Ward PB, Yung AR, Killackey E, Stubbs B. The Lancet Psychiatry Commission: a blueprint for protecting physical health in people with mental illness. Lancet Psychiatry. 2019 Aug;6(8):675-712. doi: 10.1016/S2215-0366(19)30132-4. Epub 2019 Jul 16. No abstract available. PMID 31324560
- [Background] Firth J, Solmi M, Wootton RE, Vancampfort D, Schuch FB, Hoare E, Gilbody S, Torous J, Teasdale SB, Jackson SE, Smith L, Eaton M, Jacka FN, Veronese N, Marx W, Ashdown-Franks G, Siskind D, Sarris J, Rosenbaum S, Carvalho AF, Stubbs B. A meta-review of "lifestyle psychiatry": the role of exercise, smoking, diet and sleep in the prevention and treatment of mental disorders. World Psychiatry. 2020 Oct;19(3):360-380. doi: 10.1002/wps.20773. PMID 32931092
- [Background] Suetani S, Rosenbaum S, Scott JG, Curtis J, Ward PB. Bridging the gap: What have we done and what more can we do to reduce the burden of avoidable death in people with psychotic illness? Epidemiol Psychiatr Sci. 2016 Jun;25(3):205-10. doi: 10.1017/S2045796015001043. Epub 2016 Jan 15. PMID 26768358
- [Background] Firth J, Ward PB, Stubbs B. Editorial: Lifestyle Psychiatry. Front Psychiatry. 2019 Aug 26;10:597. doi: 10.3389/fpsyt.2019.00597. eCollection 2019. No abstract available. PMID 31507466
- [Background] Hemming K, Haines TP, Chilton PJ, Girling AJ, Lilford RJ. The stepped wedge cluster randomised trial: rationale, design, analysis, and reporting. BMJ. 2015 Feb 6;350:h391. doi: 10.1136/bmj.h391. No abstract available. PMID 25662947
- [Background] Koorts H, Eakin E, Estabrooks P, Timperio A, Salmon J, Bauman A. Implementation and scale up of population physical activity interventions for clinical and community settings: the PRACTIS guide. Int J Behav Nutr Phys Act. 2018 Jun 8;15(1):51. doi: 10.1186/s12966-018-0678-0. PMID 29884236
- [Derived] van Schothorst MME, den Bleijker NM, van Harten PN, De Vries NK, Deenik J. Barriers and facilitators of inpatients and healthcare professionals prior to the implementation of a Multidisciplinary Lifestyle-Focused Approach in the Treatment of Inpatients With Mental Illness (MULTI+): The MULTI+ Study II. Implement Res Pract. 2025 Jul 6;6:26334895251351663. doi: 10.1177/26334895251351663. eCollection 2025 Jan-Dec. PMID 40630921
- [Derived] den Bleijker NM, van Schothorst MME, Hendriksen IJM, Cahn W, de Vries NK, van Harten PN, Deenik J. Effectiveness and implementation of a multidisciplinary lifestyle focused approach in the treatment of inpatients with mental illness (MULTI +): a stepped wedge study protocol. BMC Psychiatry. 2022 Mar 31;22(1):230. doi: 10.1186/s12888-022-03801-w. PMID 35361168